CLINICAL TRIAL: NCT07389590
Title: A Pilot Study of Ublituximab in People With MS Experiencing Wearing Off Phenomena While Receiving Treatment With Ocrelizumab
Brief Title: Study of Ublituximab for Ocrelizumab Wearing-Off in Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00449860
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
Keywords: wearing off; ocrelizumab; ublituximab
MeSH Terms: conditions — Multiple Sclerosis | interventions — ublituximab; ocrelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ublituximab (Experimental): Participants in this arm will switch from Ocrelizumab to receive Ublituximab administered intravenously (IV) as cumulative dose of 450-milligram (mg) infusions every 6 months for at least 2 doses.
  Interventions: Drug: Ublituximab
- Ocrelizumab (Active Comparator): Participants in this arm will continue to receive Ocrelizumab administered intravenously (IV) as 600-milligram (mg) infusions every 6 months for at least a further 2 doses.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ublituximab — Ublituzimab will be administered via IV infusion as specified throughout the study period.
  Arms: Ublituximab
Drug: Ocrelizumab — Ocrelizumab will be administered via IV infusion as specified throughout the treatment period.
  Arms: Ocrelizumab

SUMMARY:
The proposed study is a pilot study of ublituximab involving people with multiple sclerosis (MS) who are experiencing a "wearing off" phenomenon (return or worsening of MS-related symptoms) while being treated with ocrelizumab, and exploring whether switching to ublituzimab can resolve, improve or delay this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing forms of MS.
* Age between 18 and 65 years old (inclusive).
* On treatment with standard interval ocrelizumab for at least one year.
* Eligible and willing to continue treatment with ocrelizumab or ublituximab.
* The presence of wearing off phenomena, defined as either worsening in any Neuro-QoL sleep disturbance, fatigue, depression, upper and lower extremity scores (moving from a lower category of symptom severity to a higher category, based on previously defined cutoff scores), a worsening of Neuro-QoL score of 10 points (which equals 1 SD) or more in any domain between a 1-2 month post-infusion assessment (after one ocrelizumab infusion) and a 1-2 month pre-infusion assessment (before the next scheduled infusion).

Exclusion Criteria:

* Prior therapy: Has ever received any of the following:

  * B-cell targeted therapies: rituximab, ofatumumab, ublituximab or other anti-CD20 agents besides ocrelizumab.
  * Prior use of cladribine, alemtuzumab, mitoxantrone, cyclophosphamide or HSCT.
* Lymphopenia: a lymphocyte count <500/ millimeter (mm)^3. Historical labs may be used if the collection date is 6 months or less prior to deeming eligible.
* Neutrophils <1.5X10E9/L. Historical labs may be used if the collection date is 6 months or less prior to deeming eligible.
* Clinically unstable medical or psychiatric disorder.
* Substance abuse: has evidence of current drug or alcohol abuse or dependence.
* 365 Day prior therapy: has received a biologic investigational agent other than B-cell targeted therapy [e.g., anti CD40L antibody].
* Malignancy: has a history of malignancy in the past 5 years except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Have a history of a primary immunodeficiency.
* Have a significant IgG deficiency (IgG level < 400 mg/dL).
* Have an IgA deficiency (IgA level < 10 mg/dL).
* Infection history:

  * Currently on any suppressive therapy for chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria).
  * Hospitalization for treatment of infection within 60 days of Screening.
  * Use of parenteral (IV or IM) antibiotics (anti-bacterial, antiviral, anti-fungal, or anti-parasitic agents) within 60 days of Screening.
* Other disease/conditions: has any of the following: a) clinical evidence of significant unstable or uncontrolled acute or chronic diseases (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* Hepatitis status:

  * Serologic evidence of current or past Hepatitis B (HB) infection based on the results of testing for HBsAg and HBcAb as follows: Patients positive for HBsAg or HBcAb are excluded.
  * A positive test for Hepatitis C antibody
* HIV: known to have a historically positive HIV test or tests positive at screening for HIV.
* Laboratory abnormalities: An abnormal laboratory assessment is made, which is judged clinically significant by the investigator.
* Drug Sensitivity: has a history of sensitivity to any of the study medications.
* Any contraindication to undergoing MRI.
* TB: tests positive at screening for tuberculosis.
* Impaired decision-making capacity or impaired ability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients with Wearing-Off | From month 1 up to 11 months
  The proportion of patients with the wearing-off phenomenon (as defined below).
  Wearing off is defined as either worsening in any Neuro-QoL fatigue, depression, upper and lower extremity scores (moving from a lower category of symptom severity to a higher category, based on previously defined cutoff scores) or 0.5-point worsening in average SymptoMScreen score.

SECONDARY OUTCOMES:
The Frequency and Severity of Wearing-Off Events as assessed by the number of Neuro-QoL or SymptoMScreen events | From month 1 up to 11 months
  The number of Neuro-QoL or SymptoMScreen events (as defined below) per patient per infusion cycle that qualifies as a marker of wearing off.
  Wearing off events are defined as either worsening in any Neuro-QoL fatigue, depression, upper and lower extremity scores (moving from a lower category of symptom severity to a higher category, based on previously defined cutoff scores) or 0.5-point worsening in average SymptoMScreen score.

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Saidha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States